CLINICAL TRIAL: NCT00833131
Title: Short-course Preoperative Radiotherapy With Consolidating Chemotherapy vs. Preoperative Chemoradiation in Patients With Unresectable Rectal Cancer: Phase III Study
Brief Title: The Randomised Study of Preoperative Radiotherapy With Consolidating Chemotherapy for Unresectable Rectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Polish Colorectal Cancer Study Group (Network)
Collaborators: Maria Sklodowska-Curie National Research Institute of Oncology (Other); Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Cracow (Other); Poznan University of Medical Sciences (Other); Medical University of Lublin (Other)
Responsible Party: Prof. Marek P. Nowacki, Maria Sklodowska-Curie Memorial Cancer Center, Institute of Oncology in Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGBRJG0109
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2010-04

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Preoperative radiotherapy and consolidating chemotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 25 Gy in 5 fractions of 5 Gy over 5 days. One week interval. Consolidating chemotherapy of 3 courses of FOLFOX4. Surgery 10-11 weeks from beginning of radiation and at least 4 weeks from the last dose of fluorouracil.
  Interventions: Radiation: Short course of radiotherapy
- 2 (Active Comparator): Conventionally fractionated chemoradiation with 50.4 Gy total dose in 28 fractions of 1.8 Gy over 5.5 weeks. Surgery 10-11 weeks from beginning of radiation and at least 4 weeks from the last dose of radiation.
  Interventions: Radiation: Radiochemotherapy

INTERVENTIONS:
Radiation: Short course of radiotherapy — 5 x 5 Gy and afer one week interval consolidating chemotherapy of 3 courses of FOLFOX4
  Other Names: short radiation; consolidating chemotherapy
  Arms: 1
Radiation: Radiochemotherapy — 28 x 1,8 Gy with simultaneous neoadjuvant chemotherapy: two courses of 5-Fu 325 mg/m2/day i.v. bolus and LV 20 mg/m2/day i.v.-bolus over 5 days given during 1-5 and 29-33 days of radiation. Oxaliplatin is given 50 mg/m2 once a week 5 times during 1, 8, 15, 22 and 29 days of radiation.
  Other Names: chemoradiation
  Arms: 2

SUMMARY:
The addition of Oxaliplatin to conventionally fractionated chemoradiation (FULV or capecitabine) is considered as standard in unresectable rectal cancer by the panel of experts. The Investigators addressed the question whether short-course preoperative radiotherapy with consolidating chemotherapy of FOLFOX4 may increase the rate of R0 resection in patients with unresectable rectal cancer.

DETAILED DESCRIPTION:
Patients with unresectable primary rectal cancer or with unresectable local recurrence without distant metastases are randomly allocated to control or experimental arm. The preoperative treatment in the control arm is conventionally fractionated chemoradiation with 50.4 Gy total dose in 28 fractions of 1.8 Gy over 5.5 weeks simultaneously with 5-Fu, leucovorin and oxaliplatin. Experimental group receive 25 Gy in 5 fractions of 5 Gy over 5 days and after one week interval - consolidating chemotherapy of 3 courses of FOLFOX4. Surgery should be curried out 10-11 weeks from beginning of radiation and at least 4 weeks from the last dose of fluorouracil or radiation. The study hypothesis is that the short-course preoperative radiotherapy with consolidating chemotherapy produce at least 10% increase of the rate of R0 resection compared to preoperative chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable primary rectal cancer or with unresectable local recurrence without distant metastases.
* WHO performance status ≤ 2.
* Lower border of tumour ≤ 15 cm from anal verge.

Exclusion Criteria:

* cardiac coronary arterial disease,
* arrhythmias,
* stroke even if they have occurred in the past and are controlled with medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2008-11; Primary Completion 2012-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
The rate of patients with R0 resection | Surrogate endpoint available immediatly after surgery

SECONDARY OUTCOMES:
Overall long-term survival | 5 years
Progression-free long-term survival | 5 years
The rate of local failures | 5 years
The rate of distant metastases | 5 years
The rate of early toxicity of neoadjuvant treatment according to the NCI CTCAE (version 3.0) | 3 months
The rate of postoperative complications | 30 days
The rate of late toxicity according to the RTOG/EORTC scale | 5 years
The rate of complete pathological response | Surrogate endpoint available immediatly after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Bujko, Prof., Principal Investigator — Roentgena 5, 02-781 Warsaw, Poland
Locations (1):
- M. Sklodowska-Curie Memorial Cancer Centre, Warsaw, Poland

REFERENCES:
- [Background] Bujko K, Kolodziejczyk M. The 5 x 5 Gy with delayed surgery in non-resectable rectal cancer: a new treatment option. Radiother Oncol. 2008 Jun;87(3):311-3. doi: 10.1016/j.radonc.2007.12.020. Epub 2008 Jan 18. No abstract available. PMID 18207596
- [Derived] Cisel B, Pietrzak L, Michalski W, Wyrwicz L, Rutkowski A, Kosakowska E, Cencelewicz A, Spalek M, Polkowski W, Jankiewicz M, Stylinski R, Bebenek M, Kapturkiewicz B, Maciejczyk A, Sadowski J, Zygulska J, Zegarski W, Jankowski M, Las-Jankowska M, Toczko Z, Zelazowska-Omiotek U, Kepka L, Socha J, Wasilewska-Tesluk E, Markiewicz W, Kladny J, Majewski A, Kapuscinski W, Suwinski R, Bujko K; Polish Colorectal Study Group. Long-course preoperative chemoradiation versus 5 x 5 Gy and consolidation chemotherapy for clinical T4 and fixed clinical T3 rectal cancer: long-term results of the randomized Polish II study. Ann Oncol. 2019 Aug 1;30(8):1298-1303. doi: 10.1093/annonc/mdz186. PMID 31192355
- [Derived] Bujko K, Wyrwicz L, Rutkowski A, Malinowska M, Pietrzak L, Krynski J, Michalski W, Oledzki J, Kusnierz J, Zajac L, Bednarczyk M, Szczepkowski M, Tarnowski W, Kosakowska E, Zwolinski J, Winiarek M, Wisniowska K, Partycki M, Beczkowska K, Polkowski W, Stylinski R, Wierzbicki R, Bury P, Jankiewicz M, Paprota K, Lewicka M, Cisel B, Skorzewska M, Mielko J, Bebenek M, Maciejczyk A, Kapturkiewicz B, Dybko A, Hajac L, Wojnar A, Lesniak T, Zygulska J, Jantner D, Chudyba E, Zegarski W, Las-Jankowska M, Jankowski M, Kolodziejski L, Radkowski A, Zelazowska-Omiotek U, Czeremszynska B, Kepka L, Kolb-Sielecki J, Toczko Z, Fedorowicz Z, Dziki A, Danek A, Nawrocki G, Sopylo R, Markiewicz W, Kedzierawski P, Wydmanski J; Polish Colorectal Study Group. Long-course oxaliplatin-based preoperative chemoradiation versus 5 x 5 Gy and consolidation chemotherapy for cT4 or fixed cT3 rectal cancer: results of a randomized phase III study. Ann Oncol. 2016 May;27(5):834-42. doi: 10.1093/annonc/mdw062. Epub 2016 Feb 15. PMID 26884592